CLINICAL TRIAL: NCT03955445
Title: An Open-label, Non-randomized Extension Study to Evaluate the Long-term Efficacy, Safety and Tolerability of Iptacopan (LNP023) in C3 Glomerulopathy or Idiopathic Immune-complex-membranoproliferative Glomerulonephritis
Brief Title: Long-term Efficacy, Safety and Tolerability of Iptacopan in C3G or IC-MPGN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023B12001B; 2018-004253-24 (EudraCT Number); 2023-509343-27-00 (Other: EU CT Number)
Expanded Access: NCT05222412 (Available)
Record Dates: First submitted 2019-05-03; First posted 2019-05-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: C3 Glomerulopathy; Immune-complex-membranoproliferative Glomerulonephritis
Keywords: C3G; C3 glomerulopathy; C3GN; C3 glomerulonephritis; DDD; dense deposit disease; iptacopan; LNP023; IC-MPGN; idiopathic immune-complex- membranoproliferative glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: participants with native kidneys from CLNP023X2202 (Experimental): C3G participants from study CLNP023X2202 with native kidneys receiving iptacopan capsules 200 mg b.i.d
  Interventions: Drug: LNP023
- Cohort B: participants with transplanted kidneys and recurrent C3G from CLNP023X2202 (Experimental): C3G participants from study CLNP023X2202 who have undergone kidney transplant and have recurrence of C3G receiving iptacopan capsules 200 mg b.i.d
  Interventions: Drug: LNP023
- Cohort C: Participants with native C3G randomized to placebo in CLNP023B12301 (Experimental): Native C3G Participants (adults and adolescents) from CLNP023B12301 study who were randomized to placebo in the core study receiving iptacopan capsules 200mg b.i.d
  Interventions: Drug: LNP023
- Cohort D: particpants with native C3G randomised to iptacopan in CLNP023B12301 (Experimental): Native C3G participants (adults and adolescents) from study CLNP023B12301 who were randomized to iptacopan in the core study. Receiving iptacopan capsules 200mg b.i.d
  Interventions: Drug: LNP023
- Cohort E: participants with IC-MPGN randomized to placebo in CLNP023B12302 (Experimental): IC-MPGN participants (adults and adolescents) from study CLNP023B12302 who were randomized to placebo in the core study receiving iptacopan capsules 200mg b.i.d
  Interventions: Drug: LNP023
- Cohort F: participants with IC-MPGN randomized to ipatocan in CLNP023B12302 (Experimental): IC-MPGN participants (adults and adolescents) from study CLNP023B12302 who were randomized to iptacopan in the core study receiving iptacopan capsules 200mg b.i.d
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — LNP023 capsules
  Other Names: iptacopan

SUMMARY:
This is an open-label extension study to evaluate the long-term efficacy, safety and tolerability of iptacopan in subjects with C3 glomerulopathy or idiopathic immune-complex-membranoproliferative glomerulonephritis

DETAILED DESCRIPTION:
The primary purpose of this extension study is to collect long-term efficacy, safety and tolerability data in eligible participants receiving open-label iptacopan after completing treatment in the C3G Phase 2 proof of concept study CLNP023X2202.

The primary (at 9 months) and longer-term (>9 months) efficacy and safety data of iptacopan collected from CLNP023X2202 participants will be used to support health authority submissions.

This umbrella protocol will also allow:

* continued access to iptacopan to patients enrolled in the ongoing Phase 3 programs (C3G and IC-MPGN)
* C3G study (CLNP023B12301): adults and adolescents
* IC-MPGN study (CLNP023B12302): adults and adolescents
* provision of additional efficacy and safety information following longer-term treatment in C3G and IC-MPGN populations to support health authority submissions.

Efficacy and safety assessments at the 9 month visit of this extension study in combination with data from CLNP023X2202 (baseline plus 3 months of treatment) allowed evaluation of the effects of iptacopan on potential endpoint(s) at 12 months of iptacopan treatment in C3G participants. The enrollment of C3G and IC-MPGN participants (adults and adolescents) from Phase 3 studies, CLNP023B12301 and CLNP023B12302, permits longer-term evaluation of the persistence of effects observed after iptacopan treatment. These longer term efficacy and safety assessments may be compared to historical/concurrent control data available from relevant real world databases in C3G or IC-MPGN patients and used as supportive information for registration purposes.

This extension study is expected to continue until the drug product becomes commercially available and accessible (anticipated to be up to approximately 168 months from the first patient first visit date), or the benefit-risk profile is no longer positive, or the program is discontinued for business or strategic reasons.

"Baseline" refers to the Day 1 visit (pre-dose) of CLNP023X2202, CLNP023B12301 or CLNP023B12302, whereas the Day 1 visit for this C3G/IC-MPGN extension study (CLNP023B12001B) is identified as "Extension Day 1".

ELIGIBILITY:
Inclusion Criteria:

- Patients must have completed the treatment period of the CLNP023X2202, CLNP023B12301 or CLNP023B12302 study on study drug

Exclusion Criteria:

* Severe concurrent co-morbidities, e.g. advanced cardiac disease (NYHA class IV), severe pulmonary arterial hypertension (WHO class IV), or any illness or medical condition that in the opinion of the investigator and sponsor is likely to prevent the patient from safely tolerating LNP023 or complying with the requirements of the study
* Participants with an active systemic bacterial, viral or fungal infection within 14 days prior to screening, or the presence of fever ≥ 38oC (100.4oF) within 7 days prior to screening.
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for subjects
* History of HIV or any other immunodeficiency disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2036-05-30 (Estimated); Study Completion 2036-05-30 (Estimated)

PRIMARY OUTCOMES:
CLNP023X2202 Cohort A-native C3G: Number of participants who achieve the composite renal endpoint | 9-month visit
  A participant meets the requirements of the composite renal endpoint if they satisfy the following criteria at the 9-month visit in CLNP023B12001B: (1) a stable or improved eGFR compared to the baseline visit in CLNP023X2202 (≤10% reduction in eGFR), and (2) either ≥50% reduction compared to the baseline visit in CLNP023X2202 or a reduction to <300 mg/g in UPCR and (3) either a ≥50% increase in C3 compared to baseline or an increase to ≥90 mg/dL (i.e., ≥ the lower limit of normal (LLN)). Initiation of treatment with eculizumab or any other complement pathway modifying agent automatically designates the participant as not meeting the endpoint.
CLNP023X2202 Cohort B - kidney transplant and recurrent C3G: Change from baseline in the C3 Deposit Score | 6 - to 9- month visit
  Change from baseline in the C3 Deposit Score (based on immunofluorescence microscopy) compared to baseline in the CLNP023X2202 study.
Number of AEs of special interest for participants from CLNP023X2202, CLNP023B12301 and CLNP023B12302 | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Number of participants with AEs of special interest will be collected to evaluate the long-term safety and tolerability of iptacopan in participants.
Number of participants with study drug discontinuation due to an AE (or any safety issue) for participants from CLNP023X2202, CLNP023B12301 and CLNP023B12302 | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Number of participants with study drug discontinuation due to an AE to evaluate the long-term safety and tolerability of iptacopan in participants.
Number of participants with abnormal clinically significant vital signs,ECGs, and safety laboratory measurements for participants from CLNP023X2202, CLNP023B12301 and CLNP023B12302 | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Number of participants with abnormal clinically significant vital signs, ECGs, and safety laboratory measurements to evaluate the long-term safety and tolerability of iptacopan in participants.

SECONDARY OUTCOMES:
CLNP023X2202: Number of participants who achieve the 2-component composite renal endpoint | 9-month visit
  A participant is defined as achieving the composite renal endpoint if they meet the following criteria at the 9-month visit in CLNP023B12001B: (1) a stable or improved eGFR compared to the baseline visit in CLNP023X2202 (≤10% reduction in eGFR), and (2) either ≥50% reduction compared to the baseline visit in CLNP023X2202 or a reduction to <300 mg/g in UPCR.
  Initiation of treatment with eculizumab or any other complement pathway modifying agent automatically designates the participant as a not meeting the composite renal endpoint.
CLNP023X2202: Change from baseline in log-transformed urine protein/creatinine ratio (UPCR) | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Long-term effect of LNP023 on renal function in C3G subjects by assessing the change from baseline in log-transformed urine protein/creatinine ratio (UPCR)
CLNP023X2202: Change from baseline in log-transformed urine albumin/creatinine ratio (UACR) | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Long-term effect of LNP023 on renal function in C3G subjects by assessing the change from baseline in log-transformed urine albumin/creatinine ratio (UACR)
CLNP023X2202: Change from baseline in serum creatinine concentration | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Long-term effect of LNP023 on renal function in C3G subjects by assessing the change in serum creatinine compared to CLNP023X2202 baseline
CLNP023X2202: Change from baseline in estimated glomerular filtration rate (eGFR) | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Long-term effect of LNP023 on renal function in C3G subjects by assessing the change in eGFR compared to CLNP023X2202 baseline
CLNP023X2202: Status of C3G disease progression | 6 to 9 month visit
  Describe the status of C3G disease progression based on glomerular histopathology in a renal biopsy at 6 to 9 months from entry to the study compared to those obtained prior to treatment in the CLNP023X2202 study
CLNP023X2202: Log-transformed ratio to baseline in serum C3 | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Long-term effect of LNP023 on C3 by evaluating the Log-transformed ratio to baseline in serum C3
CLNP023X2202: Number of participants who achieve the composite renal endpoint | Up to 66 months
  A participant is defined as achieving the composite renal endpoint if they meet the following criteria at times >9 months in CLNP023B12001B: (1) a stable or improved eGFR compared to the baseline visit in CLNP023X2202 (≤10% reduction in eGFR), and (2) either ≥50% reduction compared to the baseline visit in CLNP023X2202 or a reduction to <300 mg/g in UPCR and (3) either a ≥50% increase in C3 compared to baseline or an increase to ≥90 mg/dL (i.e., LLN). Initiation of treatment with eculizumab or any other complement pathway modifying agent automatically designates the participant as a not meeting the composite renal endpoint.
CLNP023X2202: Plasma LNP023 concentration up to 12 months at trough | 3-months, 6-months, 9-months and 12-months visits
  Measurement of LNP023 plasma concentration to evaluate the pharmacokinetics of iptacopan in participants with prolonged treatment
CLNP023B12301 and CLNP023B12302: Change from initiation of iptacopan treatment in the core study in log-transformed UPCR over time. | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Change from initiation of iptacopan treatment in the core study in log-transformed UPCR will be assessed to evaluate the long-term effect of iptacopan on proteinuria
CLNP023B12301 and CLNP023B12302: Change from initiation of iptacopan treatment in the core study in eGFR over time. | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  Change from initiation of iptacopan treatment in the core study in eGFR over time will be assessed to evaluate the long-term effect of iptacopan on eGFR
CLNP023B12301 and CLNP023B12302: Number of participants who achieve a 2-component composite renal endpoint | Participants are expected to continue on study for a minimum of 60 months and a maximum of 84 months
  A participant is defined as meeting the requirements of the composite renal endpoint if they satisfy the eGFR (a stable or improved eGFR, i.e., ≤15% reduction in eGFR compared to the initiation of iptacopan treatment in the core study) and UPCR (≥50% reduction in UPCR compared to the initiation of iptacopan treatment in the core study) criteria assessed at a visit. Initiation of any complement pathway modifying agent or initiation/intensification of corticosteroid or immunosuppressant therapy, or renal replacement therapy automatically designates the participant as not having met the endpoint. The rate will be evaluated over time.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (5):
  - Childrens Hospital Colorado, Aurora, Colorado
  - Georgia Nephrology Research Inst, Lawrenceville, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Col Uni Med Center New York Presby, New York, New York
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Brazil (5):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Botucatu, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Novartis Investigative Site, Toronto, Ontario, Canada
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Prague, Czechia
- France (3):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (4):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Heraklion Crete., Greece
- Novartis Investigative Site, Petah Tikva, Israel
- Italy (2):
  - Novartis Investigative Site, Ranica, BG
  - Novartis Investigative Site, Roma, RM
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Niigata
- Novartis Investigative Site, Leiden, South Holland, Netherlands
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Bern, Switzerland
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Köseköy, Kocaeli
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Ankara, Yenimahalle
- United Kingdom (3):
  - Novartis Investigative Site, London, London
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Cardiff

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.